CLINICAL TRIAL: NCT04200911
Title: Cognition, Age, and RaPamycin Effectiveness - DownregulatIon of thE mTor Pathway (CARPE DIEM)
Brief Title: Cognition, Age, and RaPamycin Effectiveness - DownregulatIon of thE mTor Pathway
Acronym: CARPE_DIEM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20190850H; UL1TR002645 (NIH)
Record Dates: First submitted 2019-12-06; First posted 2019-12-16 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Cognitive Impairment, Mild; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- RAPA intervention (Experimental): Sirolimus 1mg orally once a day for 8 weeks
  Interventions: Drug: Rapamune

INTERVENTIONS:
Drug: Rapamune — Sirolimus 1mg capsules
  Other Names: Sirolimus

SUMMARY:
Evaluation of central nervous system penetration of orally administered Rapamune (RAPA) in older adults with Mild Cognitive Impairment (MCI) or early Alzheimer's disease (AD) and investigate associated safety, tolerability, target engagement, cognition, and functional status as initial proof-of-concept study

DETAILED DESCRIPTION:
This study is an open-label pilot study of orally administered RAPA to measure its target engagement in Cerebrospinal Fluid (CSF) and blood, and to establish the feasibility and safety of RAPA treatment in older adults with MCI and early stage AD as initial proof-of-concept for a larger Phase 2 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mild Cognitive Impairment (MCI) or Alzheimer's disease, Global Clinical Dementia Rating Scale (CDR)=0.5-1
* Normal blood cell counts without clinically significant excursions; ; normal liver and renal function; and glucose control (HbA1c < 6.5%). Lipid panel and PT/PTT/INR within normal limits
* A Legally Authorized Representative (LAR) if necessary for consent
* An LAR or study partner to accompany participant to all visits
* Availability for all study visits
* Stable dose of AD medications) Donepezil, rivastigmine, memantine, galantamine) for at least 3 months prior to the baseline visit

Exclusion Criteria:

* Diabetes (HbA1c≥6.5% or anti-diabetic medications)
* History of skin ulcers or poor wound healing
* Current tobacco or illicit drug use or alcohol abuse
* Use of anti-platelet or anti-coagulant medications other than aspirin
* Current medications that affect cytochrome P450 3A4; current or recent medications for hypertriglyceridemia (eg, Gemfibrozil)
* Hypersensitivity or history of allergy to Rapamycin
* Immunosuppressant therapy within the last year; current treatment with hydroxychloroquine and chloroquine (requires "washout period" of 14 days)
* Chemotherapy or radiation treatment within the last year
* Current or chronic history of liver disease or known hepatic or biliary abnormalities
* History of primary hypertriglyceridemia. Abnormal triglycerides >200 or LDL cholesterol >193, or other abnormal labs deemed clinically significant upon investigator review
* Current or chronic history of pulmonary disease or abnormal pulse oximetry (<90%)
* Chronic heart failure
* Pregnancy
* Recent history (past 6 months) of myocardial infarction, active coronary artery disease, intestinal disorders, stroke, or transient ischemic attack
* significant neurological conditions other than AD
* Poorly controlled blood pressure (systolic BP>160, diastolic BP>90mmHg)
* Active inflammatory, COVID-19, autoimmune, infectious, hepatic, gastrointestinal, malignant, and/or psychiatric disease
* History of, or Magnetic Resonance Imaging (MRI) positive for any space occupying lesion, including mass effect and/or abnormal intracranial pressure, which would indicate contraindication to lumbar puncture
* Organ transplant recipients

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitzi Gonzales, PhD, Principal Investigator — UT Health San Antonio
Locations (1):
- UTHSA McDermott Clinical Sciences Building, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The Institution, Sponsor or respective designees may review results prior to presenting or publishing the results of a scientific investigation involving this Study in accordance with ICJME guidelines and institutional requirements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication in a peer reviewed journal

REFERENCES:
- [Derived] Gonzales MM, Garbarino VR, Kautz TF, Song X, Lopez-Cruzan M, Linehan L, Van Skike CE, De Erausquin GA, Galvan V, Orr ME, Musi N, He Y, Bateman RJ, Wang CP, Seshadri S, Kraig E, Kellogg D Jr. Rapamycin treatment for Alzheimer's disease and related dementias: a pilot phase 1 clinical trial. Commun Med (Lond). 2025 May 20;5(1):189. doi: 10.1038/s43856-025-00904-9. PMID 40394335

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects that were enrolled and passed eligibility screening and went on to randomization.
Period: Overall Study
Arm/Group | RAPA Intervention
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Diagnosis [Count of Participants; unit: Participants] — Clinical diagnosis of mild cognitive impairment or early-stage Alzheimer's disease by a qualified physician
  Participants
    Mild cognitive impairment | 6
    Early-stage dementia | 4

OUTCOME MEASURES:

1. Primary Outcome: Blood Brain Barrier Penetration of RAPA
Description: Lumbar punctures will be performed at baseline and after the final RAPA dose, to assess CSF levels of the drug. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: Change from Baseline to 8 weeks
Population: HPLC/MS/MS
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
ng/ml | 0 (0)

2. Secondary Outcome: Adverse Events
Description: Number of adverse events experienced across all 10 subjects after they were enrolled and randomized to treatment, regardless of relatedness to intervention.
Time Frame: Baseline to 8 weeks
Measure: Number; unit: Events
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
Events | 20

3. Secondary Outcome: Change in Vitals From Baseline to 8 Weeks
Description: Evaluation of vitals. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: Baseline to 8 weeks
Population: paired samples t-test comparing pre to post-treatment blood pressure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
mmHg
  systolic blood pressure | 10.45 (7.82)
  diastolic blood pressure | 1.7 (5.87)

4. Secondary Outcome: Percentage of Study Drug Pills Taken
Description: Average percentage of study drug pills taken across all 10 subjects after they were enrolled and randomized to treatment. The percentage of study drug pills taken was evaluated by having participants return any leftover study drug pills at each visit during the active treatment period.
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of study drug pills taken
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
percentage of study drug pills taken | 92 (5)

5. Secondary Outcome: Change in CSF AD Biomarkers From Baseline to 8 Weeks
Description: Evaluation of CSF AD biomarkers. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: Baseline to 8 weeks
Population: paired samples t-test comparing pre to post-treatment CSF ADRD biomarker levels
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
ng/ml
  CSF ptau-181 | 2.64 (2.72)
  CSF abeta 40 | 615.57 (1210.06)
  CSF Abeta42 | 21.52 (62.12)
  CSF GFAP | 6262.21 (4928.96)
  CSF NFL | 367.18 (310.71)

6. Secondary Outcome: Change in Plasma AD Biomarkers From Baseline to 8 Weeks
Description: Evaluation of plasma AD biomarkers. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: Baseline to 8 weeks
Population: paired samples t-test comparing pre to post-treatment plasma ADRD biomarker levels
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
ng/ml
  plasma ptau-181 | -0.22 (0.47)
  plasma abeta 40 | -8.86 (12.28)
  Plasma Abeta42 | -0.67 (0.69)
  Plasma GFAP | -27.70 (64.78)
  Plasma NFL | 0.84 (4.64)

7. Secondary Outcome: Change in CSF Inflammatory Markers From Baseline to 8 Weeks
Description: Evaluation of CSF inflammatory markers. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: Baseline to 8 weeks
Population: paired samples t-test comparing pre to post-treatment CSF inflammatory values.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
pg/ml
  IL-10 | 0.02 (0.02)
  IL-6 | -0.02 (0.25)
  IL-8 | 5.76 (9.10)
  TNF-α | 0.03 (0.07)
  IL-12 | 0.35 (0.53)
  IL-15 | 0.29 (0.28)
  IL-16 | 0.63 (3.40)
  IL-17a | 0.03 (0.09)
  IL-1a | -0.15 (0.33)
  IL-5 | 0.07 (0.07)
  IL-7 | 0.004 (0.10)
  VEGF-A | 0.95 (2.37)
  VEGF-C | 266.60 (575.93)
  VEGF-D | 109.64 (117.23)
  Eotaxin | -5.05 (32.40)
  Eotaxin-3 | -0.20 (2.20)
  IP-10 | -12.93 (143.87)
  MCP-1 | -22.56 (78.00)
  MIP1-α | 0.83 (2.90)
  sFLT-1 | 41.18 (253.61)
  PIGF | 2.84 (40.66)
  bFGF | -0.69 (20.85)
  sVCAM1 | 21202.57 (24439.62)
  sICAM1 | 6701.21 (13402.98)
  SAA | -73762.91 (375497.74)
  CRP | -98910.45 (27540.81)
  IFN-γ | 0.14 (0.17)

8. Secondary Outcome: Change in Plasma Inflammatory Markers From Baseline to 8 Weeks
Description: Evaluation of plasma inflammatory markers. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: Baseline to 8 weeks
Population: paired samples t-test comparing pre to post-treatment plasma inflammatory biomarkers.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
pg/ml
  IL-10 | -0.18 (0.53)
  IL-6 | 0.29 (0.54)
  IL-8 | 0.16 (1.57)
  TNF-α | 0.06 (0.44)
  IL-12 | -16.56 (38.52)
  IL-15 | 0.12 (0.31)
  IL-16 | 16.18 (42.70)
  IL-17a | 0.36 (1.68)
  IL-1a | -0.20 (0.36)
  IL-5 | 0.34 (0.46)
  IL-7 | -0.14 (1.63)
  VEGF-A | -0.05 (7.98)
  VEGF-C | 2000.38 (6648.40)
  VEGF-D | 3741.02 (3124.38)
  Eotaxin | 22.07 (36.04)
  Eotaxin-3 | -3.60 (6.19)
  IP-10 | 18.26 (80.08)
  MCP-1 | -4.80 (10.74)
  MIP1-α | -0.83 (3.64)
  sFLT-1 | 258.88 (237.44)
  PIGF | 20.81 (11.81)
  bFGF | -143.67 (174.71)
  sVCAM1 | 97456.61 (1400309.82)
  sICAM1 | 91844.33 (1329185.57)
  SAA | 190090000 (936172849.0)
  CRP | 36165816.2 (111516450.7)
  IFN-γ | 4.37 (1.91)

9. Secondary Outcome: Safety Labs - Change in White Blood Cell and Platelet Counts From Baseline to 8 Weeks
Description: Evaluation of safety labs - white blood cell and platelet counts. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: Baseline to 8 weeks
Population: paired samples t-test comparing pre to post-treatment safety laboratory values.
Measure: Mean (Standard Deviation); unit: x10^3 cells/μL
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
x10^3 cells/μL
  White Blood Cell Count | 0.42 (1.92)
  Immature Granulocytes | -0.21 (1.19)
  Eosinophils | 0.10 (2.5)
  Basophils | -0.19 (0.40)
  Platelets | 20.60 (35.19)

10. Secondary Outcome: Safety Labs - Change in Red Blood Cell Count
Description: Evaluation of safety labs - red blood cell counts. Change in red blood cell count calculated as value at 8 weeks minus the value at baseline.
Time Frame: Baseline to 8 weeks
Population: paired sample's t-test comparing pre to post-treatment safety laboratory values
Measure: Mean (Standard Deviation); unit: x10^6 cells/μL
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
x10^6 cells/μL | -0.01 (0.27)

11. Secondary Outcome: Safety Labs - Change in Mean Corpuscular Volume
Description: Evaluation of safety labs - Change in Mean Corpuscular volume. Change is calculated as value at 8 weeks minus the value at baseline
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
fL | -2.70 (2.16)

12. Secondary Outcome: Safety Labs - Change in Mean Corpuscular Hemoglobin
Description: safety labs - Mean Corpuscular Hemoglobin. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8-weeks
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
pg | -0.81 (0.69)

13. Secondary Outcome: Safety Labs - Change in Metabolic Parameters (g/dl)
Description: Evaluation of safety labs - metabolic parameters. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
g/dl
  Hemoglobin | -0.27 (0.57)
  Protein | -1.77 (5.85)
  Albumin | -0.13 (0.19)
  Mean Corpuscular Hemoglobin Concentration | 0.08 (0.85)

14. Secondary Outcome: Safety Labs - Change in Hematocrit
Description: Evaluation of of safety labs - hematocrit. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
percentage of red blood cells | -0.86 (2.09)

15. Secondary Outcome: Safety Labs - Change in Monocytes
Description: Evaluation of of safety labs - monocytes. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of white blood cell count
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
percentage of white blood cell count | -0.19 (4.08)

16. Secondary Outcome: Safety Labs - Change in Red Cell Distribution Width
Description: Evaluation of of safety labs - Red cell distribution width. Change is calculated as value at 8 weeks minus the value at baseline. The value reported is % of red blood cell size and volume variability.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
Percentage | -0.65 (0.24)

17. Secondary Outcome: Safety Labs - Change in Hemoglobin A1c
Description: Evaluation of of safety labs - hemoglobin A1c. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: % of hemoglobin covered w/ glucose
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
% of hemoglobin covered w/ glucose | 0.17 (0.22)

18. Secondary Outcome: Safety Labs - Change in Metabolic and Lipid Parameters (mg/dl)
Description: Evaluation of safety labs - metabolic and lipid parameters. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
mg/dl
  glucose | 2.70 (6.67)
  blood urea nitrogen | -1.80 (4.13)
  Creatinine | -0.001 (0.09)
  Bilirubin | -0.09 (0.34)
  Cholesterol | -0.30 (26.08)
  High-Density Lipoprotein Cholesterol | 2.90 (7.22)
  Low-Density Lipoprotein Cholesterol | -2.70 (20.38)
  Very Low-Density Lipoprotein Cholesterol | -0.50 (4.25)

19. Secondary Outcome: Safety Labs - Change in Sodium and Potassium (mmol/L)
Description: Evaluation of safety labs - sodium and potassium. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
mmol/L
  Sodium | -5.40 (18.90)
  Potassium | -0.19 (0.44)

20. Secondary Outcome: Safety Labs - Change in Liver Panel (iU/L)
Description: Evaluation of safety labs - liver panel. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
IU/L
  Aspartate Aminotransferase | 1.00 (4.06)
  Alanine Transaminase | 0.001 (6.20)
  Alkaline Phosphatase | 4.10 (10.90)

21. Secondary Outcome: Cognition/Functional Status - Change in Montreal Cognitive Assessment (MoCA)
Description: The Montreal Cognitive Assessment (MoCA) assesses global cognition with scores ranging from 0 to 30 points. Higher scores indicate better performance.Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | -1.30 (2.45)

22. Secondary Outcome: Cognition/Functional Status - Change on the Clinical Rating Scale Global Score
Description: The Clinical Rating Scale Global Score assesses cognition and daily functioning with scores ranging from 0 to 3 points. Higher scores indicate worse cognition and/or functional status.Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | 0.15 (0.16)

23. Secondary Outcome: Cognition/Functional Status - Change on the Clinical Rating Scale Sum of Boxes Score
Description: The Clinical Rating Scale Sum of Boxes assesses cognition and daily functioning with scores ranging from 0 to 18 points. Higher scores indicate worse cognition and/or functional status.Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | 0.55 (0.86)

24. Secondary Outcome: Cognition/Functional Status - Change on the Hopkins Verbal Learning Test - Revised Immediate Recall
Description: The Hopkins Verbal Learning Test - Revised Immediate Recall assesses verbal list learning with scores ranging from 0 to 36 points. Higher scores indicate better performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | 0.40 (3.37)

25. Secondary Outcome: Cognition/Functional Status - Change on the Hopkins Verbal Learning Test - Revised Delayed Recall
Description: The Hopkins Verbal Learning Test - Revised Delayed Recall assesses verbal list learning with scores ranging from 0 to 12 points. Higher scores indicate better performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | -1.00 (2.54)

26. Secondary Outcome: Cognition/Functional Status - Change on the Craft Story Immediate Recall Verbatim
Description: The Craft Story Immediate Recall Verbatim assesses verbal narrative learning with scores ranging from 0 to 44 points. Higher scores indicate better performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | 0.20 (4.29)

27. Secondary Outcome: Cognition/Functional Status - Change on the Craft Story Delayed Recall Verbatim
Description: The Craft Story Delayed Recall Verbatim assesses verbal memory recall with scores ranging from 0 to 44 points. Higher scores indicate better performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | -1.40 (2.95)

28. Secondary Outcome: Cognition/Functional Status - Change on the Benson Figure Copy
Description: The Benson Figure Copy assesses visuoconstructional skills with scores ranging from 0 to 17points. Higher scores indicate better performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | 0.70 (1.83)

29. Secondary Outcome: Cognition/Functional Status - Change on the Benson Figure Delayed Recall
Description: The Benson Figure Delayed Recall assesses visual memory with scores ranging from 0 to 17 points. Higher scores indicate better performance.Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | -0.80 (2.04)

30. Secondary Outcome: Cognition/Functional Status - Change on the Number Span Forward
Description: The Number Span Forward test assesses basic attention with scores ranging from 0 to 16 points. Higher scores indicate better performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | 0.20 (1.62)

31. Secondary Outcome: Cognition/Functional Status - Change on the Number Span Backward
Description: The Number Span Backward test assesses working memory with scores ranging from 0 to 14 points. Higher scores indicate better performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | -0.60 (0.84)

32. Secondary Outcome: Cognition/Functional Status - Change on the Trail Making Test Part A, Time to Completion
Description: The Trail Making Test Part A, time to completion assesses psychomotor speed and visual scanning with scores ranging from 1 to 150 seconds. Higher scores indicate worse performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: seconds to complete
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
seconds to complete | 3.09 (3.15)

33. Secondary Outcome: Cognition/Functional Status - Change Trail Making Test Part B, Time to Completion
Description: The Trail Making Test Part B, time to completion assesses attentional shifting with scores ranging from 1 to 300 seconds. Higher scores indicate worse performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: seconds to complete
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
seconds to complete | 26.69 (14.97)

34. Secondary Outcome: Cognition/Functional Status - Change on Phonemic Fluency
Description: The Phonemic fluency test assesses speeded word generation to a phonemic cue. Scores begin at 0 with no upper limit. Higher scores indicate better performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | 1.80 (3.71)

35. Secondary Outcome: Cognition/Functional Status - Change on Semantic Fluency
Description: The Semantic fluency test assesses speeded word generation to a semantic cue. Scores begin at 0 with no upper limit. Higher scores indicate better performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | 1.10 (4.18)

36. Secondary Outcome: Cognition/Functional Status - Change on the Multilingual Naming Test
Description: The Multilingual Naming Test assesses confrontation naming. Scores range from 0 to 32 and higher scores indicate better performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | 1.50 (4.67)

37. Secondary Outcome: Cognition/Functional Status - Change on the Hayling, Total Errors
Description: The Hayling assesses response inhibition errors. Scores range from 0 to 30 and higher scores indicate worse performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | 0.001 (0.78)

38. Secondary Outcome: Cognition/Functional Status - Change on Grip Strength, Dominant Hand
Description: The grip strength, dominant hand assesses grip strength in kilograms. Values begin at 0 with no upper limit. Higher scores indicate better performance Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
kilograms | 0.30 (2.10)

39. Secondary Outcome: Cognition/Functional Status - Change on Grip Strength, Non-dominant Hand
Description: The grip strength, non-dominant hand assesses grip strength in kilograms. Values begin at 0 with no upper limit. Higher scores indicate better performance. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
kilograms | -0.25 (3.30)

40. Secondary Outcome: Cognition/Functional Status - Change on the Geriatric Depression Scale 15-item
Description: The Geriatric Depression Scale 15-item assesses depressive symptomatology. Scores range from 0 to 15 and higher scores indicate worse outcomes. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | 0.10 (1.73)

41. Secondary Outcome: Cognition/Functional Status - Change on the Functional Activities Questionnaire
Description: The Functional Activities Questionnaire assesses functional status for independent activities of daily living. Scores range from 0 to 30 and higher scores indicate worse outcomes. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | -0.10 (4.36)

42. Secondary Outcome: Cognition/Functional Status - Change on the Neuropsychiatric Inventory Questionnaire
Description: The Neuropsychiatric Inventory Questionnaire assesses neuropsychiatric symptoms. Scores range from 0 to 12 and higher scores indicate worse outcomes. Change is calculated as value at 8 weeks minus the value at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RAPA Intervention
Number analyzed (Participants) | 10
score on a scale | 0.70 (2.83)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: All adverse events that occurred after enrollment and randomization are reported, whether considered not related to or possible related to intervention.
Arm/Group | RAPA Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAPA Intervention (N=10)
Altered Mental Status (Nervous system disorders) | 1 (1) — Unrelated to study intervention, possible TIA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAPA Intervention (N=10)
Intermittent Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Mild and unlikely to be related to intervention
Headache (Nervous system disorders) | 1 (1) — Moderate and not related to intervention
Urinary retention (Renal and urinary disorders) | 1 (1) — Mild and unlikely related to intervention
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1) — Mild and unlikely to be related to intervention
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Mild and unlikely to be related to intervention for one subject, possible for the other
Skin infection (Skin and subcutaneous tissue disorders) | 1 (2) — Not related to intervention (kitten scratches)
Leg edema (Blood and lymphatic system disorders) | 2 (2) — Mild for one subject, moderate for the other and unlikely to be related to intervention
Emesis (Gastrointestinal disorders) | 1 (2) — Mild, unlikely to have been related to study intervention
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Mild and not likely to be related to intervention
Diarrhea (Gastrointestinal disorders) | 1 (2) — Mild, one subject was possibly related, the other was not
Urinary incontinence (Renal and urinary disorders) | 1 (1) — Mild and unlikely related
Urinary urgency (Renal and urinary disorders) | 1 (1) — Mild and unlikely related
Fall (General disorders) | 2 (2) — Mild and unlikely related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT04200911/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT04200911/ICF_001.pdf